CLINICAL TRIAL: NCT07085039
Title: A Phase II, Single-Arm Open-Label Multi-Center Study of Ruxolitinib in Previously Treated Idiopathic Multicentric Castleman Disease
Brief Title: Ruxolitinib in Previously Treated Idiopathic Multicentric Castleman Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Incyte Corporation (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 858269
Record Dates: First submitted 2025-05-20; First posted 2025-07-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Castleman's Disease (CD); Idiopathic Multicentric Castleman's Disease
MeSH Terms: conditions — Castleman Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ruxolitinib (Other): This is an open-label study so all patients will be assigned to the same interventional arm and given ruxolitinib
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Participants will take the study drug in a tablet form, by mouth, every day for the next year, as long as it is helping with their disease and not causing unacceptable side effects.

SUMMARY:
The research study is being done to look at the effects of ruxolitinib in adults with idiopathic Multicentric Castleman Disease (iMCD) that has not gotten better from taking siltuximab or tocilizumab, or who cannot take those medications.

DETAILED DESCRIPTION:
There is currently no agreed-on recommended treatment for iMCD patients whose disease does not respond to siltuximab or tocilizumab, which is a major challenge for patients. The purpose of this study is to find out the effects of a study drug, ruxolitinib (also called Jakafi), in these patients. This study looks at how well the drug is tolerated by participants and its effects on participants' iMCD symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-80
2. Documented disease history consistent with diagnostic criteria for iMCD

   • Indication of clinico-histopathological features consistent with iMCD as determined by a licensed pathologist in a diagnostic pathology report, or a CAS grade of at least 3 in the companion registry study (ACCELERATE).
3. Refractory (patient did not achieve sufficient disease control with anti-IL-6 therapy, as determined by the site investigator), relapsed (return of symptoms while on therapy), or inability to tolerate anti-IL-6 or anti-IL-6 receptor therapy
4. Evidence of active disease, defined by at least two of: constitutional symptoms (fatigue, night sweats, fever, weight change), hemoglobin < lower limit of normal, C-reactive protein > upper limit of normal (or >10 mg/L), or albumin < lower limit of normal (<3.5 g/dL), at lease one lymph node meeting modified Cheson criteria
5. Ability to consume oral medication in the form of a tablet
6. Ability to provide informed consent prior to any study-specific activities

Exclusion Criteria:

1. Subjects cannot be pregnant or nursing females

   • Women of childbearing potential must have a negative pregnancy test documented at the Baseline Visit. Subjects of reproductive potential may not participate unless they have agreed, as part of the informed consent, to use an effective contraceptive method for the duration of the study and for at least 12 weeks after ending treatment
2. Subjects cannot have received any systemic therapy(ies) intended to treat iMCD other than corticosteroids or anti-IL-6 therapy within 14 days of enrollment

   • Corticosteroid treatment must have been initiated more than 28 days prior to enrollment and be maintained at a stable or tapering dose (prednisone or equivalent up to 1 mg/kg/day) prior to enrollment; dose cannot be elevated for the duration of the study but can be maintained or tapered

   • For subjects who cannot or are unwilling to undergo a 14-day washout period from their anti-IL-6 therapy: i. Anti-IL-6 therapy may be permitted if the subject has been on therapy for at least 3 months, no toxicity has been documented, and sufficient disease control is not achieved ii. Anti-IL-6 therapy is recommended to be discontinued within the first 6 weeks after starting ruxolitinib
3. Subjects cannot have previously received ruxolitinib monotherapy or combination therapy to treat iMCD
4. Subjects cannot have uncontrolled infection or infectious disease(s) that is/are exclusionary for / mimickers of iMCD

   * Fungal disease must be stable for at least two weeks before enrollment
   * Subjects with history of recent bacteremia must have a documented negative blood culture before enrollment
   * Subjects with past history of non-therapy related opportunistic infection should discuss eligibility and possible immunologic evaluation with the licensed site investigator prior to enrollment
5. Subjects cannot have:

   * ECOG >3
   * eGFR <30mL/min/1.73 m2 or creatinine >3.0 mg/dL
   * Absolute neutrophil count (ANC) < 1000 x 109/L
   * Hemoglobin ≤ 6.5 g/dL (transfusion independent, defined as not receiving a red blood cell transfusion for ≥ 7 days prior)
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) laboratory values greater than three times the upper limit of normal
   * Albumin < 2 g/dL (transfusion independent, defined as not receiving intravenous albumin for ≥ 7 days prior)
   * Platelet count ≤ 40 x 109/L (transfusion independent, defined as not receiving platelet transfusion for ≥ 7 days prior)
   * Pulmonary involvement or interstitial pneumonitis with dyspnea (adequate pulmonary function is defined as pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest, history of interstitial pneumonitis, etc.)
   * Fasting cholesterol > 300 mg/dL or fasting triglyceride > 400 mg/dL
6. Subjects cannot have rheumatologic disease(s) that is/are exclusionary for / mimickers of iMCD
7. Subjects cannot have a prior malignancy except for: (1) adequately treated basal cell or squamous cell skin cancer, (2) in situ cervical cancer, or (3) other cancer for which the subject has not received treatment within one year prior to enrollment

   • Other cancers will only be acceptable if the patient's life expectancy exceeds five years and they are not exclusionary diagnoses for iMCD
8. Subjects cannot have a documented history of human immunodeficiency virus (HIV) or HHV-8 infection, or severe combined immunodeficiency syndrome
9. Subjects cannot have active infections of mycobacterium tuberculosis, hepatitis B, or hepatitis C due to the potential reactivation with ruxolitinib

   * A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antigen (HBsAb) positive and hepatitis B core antibody (HBcAb) negative), or a fully resolved acute hepatitis B infection is not an exclusion criterion.
   * Subjects with an indolent chronic hepatitis B infection (normal ALT, AST, albumin and no radiographic or biopsy evidence of cirrhosis) may be eligible.
   * Subjects with active hepatitis C are excluded. Subjects positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
10. Subjects cannot have had any major adverse cardiac events, including ischemic stroke and myocardial infarction, within 6 months of enrollment
11. Subjects cannot have ongoing or planned participation in another clinical trial involving iMCD directed treatment or that involves immunomodulatory or anti-neoplastic treatment
12. Subjects cannot have prior sensitivity / allergy to any formulation of ruxolitinib, its components, or its analogues
13. Subjects cannot have serious medical illness, or psychiatric illness or disorders that could potentially interfere with the completion of treatment according to this protocol or participation in the trial
14. Subjects cannot have psychiatric disorders that compromise their ability to provide informed consent
15. Subjects cannot have any other condition or finding that, in the opinion of the investigator, would make participation in this trial inappropriate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants achieving a positive Clinical Benefit Response (CBR) response at 12 months ± 1 month. Assessments at 12 months ± 1 month. will be compared to those at the baseline visit | 12 months ± 1 month
  Clinical Benefit Response (CBR):CBR is defined by improvements in clinical symptoms (fatigue, anorexia, fever and night sweats). Laboratory markers like Hemoglobin levels, weight change and lymph node size are included in the CBR. A CBR is considered positive if there is at least a 25% reduction in the size of the largest lymph node (measured by modified Cheson criteria), a significant improvement in at least one laboratory marker (e.g., hemoglobin), and improvement in at least one clinical symptom without worsening of others.
  Positive response: Relative to baseline, improvement in at least one of the criterion without worsening of any single criterion other than hemoglobin on two consecutive study visits.
  Negative response: Relative to baseline, worsening of any single criterion other than hemoglobin on two consecutive site visits or failure to achieve improvement for any criterion.

SECONDARY OUTCOMES:
The proportion of participants achieving a positive CBR response at 3, 6, 9 months compared to baseline | 3, 6, and 9 months compared to baseline
  Clinical Benefit Response (CBR):CBR is defined by improvements in clinical symptoms (fatigue, anorexia, fever and night sweats). Laboratory markers like Hemoglobin levels, weight change and lymph node size are included in the CBR. A CBR is considered positive if there is at least a 25% reduction in the size of the largest lymph node (measured by modified Cheson criteria), a significant improvement in at least one laboratory marker (e.g., hemoglobin), and improvement in at least one clinical symptom without worsening of others
Disease activity, as measured by the CHAP scale, at 3, 6, 9, and 12 months ± 1 month. Assessments will be compared to those obtained at the Baseline Visit | 3, 6, 9, and 12 months ± 1 month
  The CHAP scale, which integrates C-reactive protein (CRP), hemoglobin, albumin levels, and Eastern Cooperative Oncology Group (ECOG) performance status, will be used to assess overall disease activity. CHAP is made up of four scores that are rated from 0-4. The sum of the four scores provides an objective scale for measuring a patient's disease activity and monitoring how it changes over time. The scale range is 0-16. A reduction in CHAP scores indicated decreased disease activity. A higher score indicates greater disease activity.
Disease activity, as measured by MCD-related Overall Symptom Score as measured by 34 outcome measures at 3, 6, 9, and 12 months ± 1 month compared to those obtained at the Baseline Visit | 3, 6, 9, and 12 months ± 1 month
  MCD-related Overall Symptom Score is measured by 34 MCD-related outcome measures. The Overall Symptom Score, comprising 34 outcome measures (fatigue, weight change, night sweats, etc.), will be used to evaluate the broader impact of Ruxolitinib on disease symptoms.
The proportion of participants achieving a lymph node response, following the modified Cheson response criteria compared to baseline | Month 12
  Radiological response will be assessed using the modified Cheson criteria, which quantifies changes in lymph node size. A lymph node response was defined as a 25% reduction in bi-dimensional measurements of the largest lymph node compared to baseline
The proportion of participants that remain on study drug for the duration of the study | Up to 73 weeks
  Number of patients who remained on the study drug for the entire study
The proportion of participants that indicate that they are currently receiving Ruxolitinib at the end of the Follow-Up Phase | Up to 73 weeks
  Number of participants who continue to take the drug until the end of the follow up phase

OTHER OUTCOMES:
All serious adverse events (SAEs) or Grade 3 or higher adverse events (AEs) related to ruxolitinib will be assessed. | 12 months
  Severe adverse events will be assessed to evaluate if there are any new, serious risks of using ruxolitinib in the iMCD population, given that ruxolitinib already has an established safety profile. AEs rated as severity level Grade 3 or higher (or moderate or higher if not in CTCAE v5) per the CTCAE v5 severity rating criteria occurring during the study period (from the time of first dosing through final visit) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: David Fajgenbaum, MD, MBA, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing may be considered upon reasonable request to the Principal Investigator, with appropriate agreements in place